CLINICAL TRIAL: NCT00036192
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of FK614 in Type 2 Diabetics Inadequately Controlled on a Sulfonylurea
Brief Title: Trial of FK614 in Type 2 Diabetics Inadequately Controlled on a Sulfonylurea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FA-614-0004
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: FK614

SUMMARY:
The purpose of the study is to assess the safety and efficacy of FK614 in type 2 diabetic subjects receiving sulfonylurea (SU) monotherapy.

DETAILED DESCRIPTION:
This is a prospective randomized, double-blind, placebo controlled, parallel group, Phase 2 study. Subjects meeting selection criteria will be randomly assigned to receive 12 weeks twice daily (BID) dosing with FK614 or placebo. Enrollment for this study will be approximately 200 patients.

ELIGIBILITY:
Inclusion Criteria

* Has history of type 2 diabetes mellitus for at least 1 year
* Has been taking current sulfonylurea (SU) for at least 3 months. Subjects currently taking metformin may be eligible to be switched.
* Has not received any oral antidiabetic medication other than an SU or taken regularly prescribed insulin for at least 3 months

Exclusion Criteria

* Has type 1 diabetes mellitus
* Has uncontrolled hypertension, i.e., systolic BP >170 or diastolic BP > 95 mm Hg.
* History of congestive heart failure

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-02; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - International Institute of Clinical Research, Inc., Ozark, Alabama
  - Arizona Research Associates, Tucson, Arizona
  - OCCR @ East Gate Medical Center, Cypress, California
  - Clinical Trials of St. Jude Heritage Md Grp, Fullerton, California
  - Research Foundation of America, Los Angeles, California
  - Progressive Clinical Research, Vista, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Physician's Office, Miami, Florida
  - University of Miami, Diabetes Center, Miami, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Central Florida Clinical Studies, Ocoee, Florida
  - Clireco, Inc., Tamarac, Florida
  - The Emory Clinic, Atlanta, Georgia
  - East-West Medical Institute, Honolulu, Hawaii
  - McConnehey Family Medicine, Nampa, Idaho
  - Physician's Office, Peoria, Illinois
  - Clinical Research, Inc., Waltham, Massachusetts
  - Radiant Research - Minneapolis, Edina, Minnesota
  - Physician's East, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Radiant Research, Mogadorf, Ohio
  - Physician's Office, Portland, Oregon
  - Physicians for Clinical Research, Camp Hill, Pennsylvania
  - Fleetwood Medical Associates, Fleetwood, Pennsylvania
  - Founders Research Corp., Philadelphia, Pennsylvania
  - SFM Clinical Trials, Scotland, Pennsylvania
  - Heartland Medical PC, New Tazewell, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Mercury Research, Inc., Houston, Texas
  - Diabetes / Glandular Disease Research Associates, San Antonio, Texas
  - Sam Clinical Research Center, San Antonio, Texas
  - McGuire Research Institute, Richmond, Virginia
  - Physician's Office, Spokane, Washington
  - University Physicians Internal Medicine, Huntington, West Virginia